CLINICAL TRIAL: NCT00959660
Title: Study of the Effect of Caloric Restriction and Exercise Training in Patients With Heart Failure and a Normal Ejection Fraction.(SECRET)
Brief Title: Exercise Intolerance in Elderly Patients With Diastolic Heart Failure
Acronym: SECRET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00005668; R37AG018915 (NIH)
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2018-04-11 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure, Diastolic; Obesity
Keywords: Diastolic heart failure; Heart Failure; Elderly; Obesity
MeSH Terms: conditions — Heart Failure, Diastolic; Obesity; Heart Failure | interventions — Exercise; Diet Therapy; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise Training (Active Comparator): Exercise participants will undergo a 1-hour supervised exercise program 3 times per week for 20 weeks consisting primarily of walking exercise using an individualized exercise prescription based on the initial exercise stress testing results.
  Interventions: Behavioral: Exercise
- Dietary Intervention (Active Comparator): A hypocaloric diet will be developed to achieve a 2800 kcal/week deficit, which should produce about 0.4 kg (1 lb) weight loss per week.
  Interventions: Dietary Supplement: Dietary Intervention
- Attention control (Active Comparator): Attention control participants will be provided a counseling session regarding general health education at baseline and will be contacted by staff via telephone every 2 weeks to discuss general health status.
  Interventions: Other: Attention Control
- Diet and Exercise (Active Comparator): A hypocaloric diet will be developed to achieve a 2450 kcal/week deficit in addition to undergoing a 1-hour supervised exercise program 3 times per week for 20 weeks consisting primarily of walking exercise using an individualized exercise prescription based on the initial exercise stress testing results.
  Interventions: Behavioral: Exercise; Behavioral: Diet and exercise

INTERVENTIONS:
Behavioral: Exercise — walking, treadmill and bicycle exercise
  Arms: Diet and Exercise; Exercise Training
Dietary Supplement: Dietary Intervention — Subjects will be provided meals and instructions for individual food selections.
  Arms: Dietary Intervention
Behavioral: Diet and exercise — Subjects will be provided meals and instructions for individual food selections and will undergo walking, treadmill and bicycle exercise.
  Arms: Diet and Exercise
Other: Attention Control — control group- continue their previously randomized life style
  Arms: Attention control

SUMMARY:
The purpose of this study is to examine the effects of weight loss via hypocaloric diet, aerobic exercise training, combined hypocaloric diet and exercise training, and attention control in patients with heart failure and a normal ejection fraction (HFNEF) and body mass index greater than or equal to 30.

DETAILED DESCRIPTION:
Heart failure with a normal ejection fraction (HFNEF, previously termed diastolic heart failure), accounts for the majority of heart failure cases in the population > 65 years old and has been recognized as a true geriatric syndrome. Exercise intolerance is the primary chronic symptom of HFNEF and a major determinant of these patients' severely reduced quality of life; however little is known regarding its pathophysiology and treatment. Therefore, our work has focused on understanding the pathophysiology of exercise intolerance in HFNEF and developing and testing interventions that may improve this pivotal outcome in this highly prevalent disorder of older persons. The aims of the proposed study are to conduct a randomized, controlled, single-blinded, 2x2 design trial to examine the effects of weight loss via hypocaloric diet, aerobic exercise training, combined hypocaloric diet and exercise training, and attention control in patients with HFNEF and body mass index >30 in order to test the following hypotheses: 1) Both weight loss and exercise training will improve exercise intolerance and quality of life in older, obese patients with HFNEF; 2) The combination of weight loss and exercise training will produce complementary effects on body and thigh muscle composition and additive improvements in exercise intolerance in HFNEF; 3) Improvements in exercise intolerance will correlate with improvements in lean body mass, reversal of adverse thigh muscle remodeling, and increased thigh muscle capillarity. The study has the potential to significantly advance our understanding of exercise intolerance and its treatment in the large population of older persons with HFNEF.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure clinical score greater than or equal to 3
* Age 60 and over
* Normal ejection fraction greater than or equal to 50%
* BMI greater than or equal to 30

Exclusion Criteria:

* Valvular heart disease
* Significant change in cardiac medication <4 weeks
* Uncontrolled hypertension
* Recent or debilitating stroke
* Cancer or other noncardiovascular conditions with life expectancy less than 2 years
* Significant Anemia
* Renal insufficiency (creatinine >2.5mg/dl)
* Psychiatric disease- uncontrolled major psychoses, depressions, dementia, or personality disorder
* Plans to leave area within 6 months
* Refuses informed consent
* Failure to pass screening test:pulmonary function, echocardiogram,or exercise

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2012-08-15 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W Kitzman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Singleton MJ, Nelson MB, Samuel TJ, Kitzman DW, Brubaker P, Haykowsky MJ, Upadhya B, Chen H, Nelson MD. Left Atrial Stiffness Index Independently Predicts Exercise Intolerance and Quality of Life in Older, Obese Patients With Heart Failure With Preserved Ejection Fraction. J Card Fail. 2022 Apr;28(4):567-575. doi: 10.1016/j.cardfail.2021.10.010. Epub 2021 Nov 10. PMID 34774747
- [Derived] Anderson T, Cascino TM, Koelling TM, Perry D, Grafton G, Houston DK, Upadhya B, Kitzman DW, Hummel SL. Measured Versus Estimated Resting Metabolic Rate in Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2021 Aug;14(8):e007962. doi: 10.1161/CIRCHEARTFAILURE.120.007962. Epub 2021 Aug 4. PMID 34344169
- [Derived] Haykowsky MJ, Nicklas BJ, Brubaker PH, Hundley WG, Brinkley TE, Upadhya B, Becton JT, Nelson MD, Chen H, Kitzman DW. Regional Adipose Distribution and its Relationship to Exercise Intolerance in Older Obese Patients Who Have Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2018 Aug;6(8):640-649. doi: 10.1016/j.jchf.2018.06.002. Epub 2018 Jul 11. PMID 30007558
- [Derived] Maldonado-Martin S, Brubaker PH, Eggebeen J, Stewart KP, Kitzman DW. Association Between 6-Minute Walk Test Distance and Objective Variables of Functional Capacity After Exercise Training in Elderly Heart Failure Patients With Preserved Ejection Fraction: A Randomized Exercise Trial. Arch Phys Med Rehabil. 2017 Mar;98(3):600-603. doi: 10.1016/j.apmr.2016.08.481. Epub 2016 Sep 28. PMID 27693420
- [Derived] Kitzman DW, Brubaker P, Morgan T, Haykowsky M, Hundley G, Kraus WE, Eggebeen J, Nicklas BJ. Effect of Caloric Restriction or Aerobic Exercise Training on Peak Oxygen Consumption and Quality of Life in Obese Older Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2016 Jan 5;315(1):36-46. doi: 10.1001/jama.2015.17346. PMID 26746456

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Training: Based on initial evaluations and the stress testing results, (HR(heart rate), VO2(maximal volume of oxygen that the body can deliver to the working muscles per minute), RPE(rate perceived exertion) an individualized exercise prescription will be developed for each subject.
  Exercise: walking, treadmill and bicycle exercise
- Diet and Exercise: The diet and exercise group is a combination of the two groups previously described.
  Exercise: walking, treadmill and bicycle exercise
  Diet and exercise: Combination of the exercise and diet group as previously described.
Period: Overall Study
Arm/Group | Exercise Training | Dietary Intervention | Attention Control | Diet and Exercise
Started | 26 | 24 | 25 | 25
Completed | 24 | 24 | 22 | 22
Not Completed | 2 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Training | Dietary Intervention | Attention Control | Diet and Exercise | Total
Number analyzed (Participants) | 26 | 24 | 25 | 25 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (5.9) | 66.5 (4.9) | 65.6 (4.8) | 66.3 (5.2) | 66.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 20 | 20 | 81
  Male | 5 | 4 | 5 | 5 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 13 | 9 | 12 | 45
  White | 15 | 11 | 16 | 13 | 55
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Exercise Capacity
Description: Exercise capacity assessed as Peak VO2 (ml/kg/min) via treadmill cardiopulmonary exercise testing using the modified Naughton protocol to the end point of exhaustion.
Time Frame: 20 weeks
Measure: Mean (95% Confidence Interval); unit: ml/kg/min
Arm/Group | Exercise Training | Dietary Intervention | Attention Control | Diet and Exercise
Number analyzed (Participants) | 24 | 24 | 22 | 22
ml/kg/min | 15.5 [15.1 to 15.9] | 15.5 [15.1 to 15.9] | 14.1 [13.5 to 14.7] | 16.6 [16.0 to 17.2]
Statistical Analysis 1: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Test type: Superiority; p < 0.001, ANCOVA — Main effects analysis with Diet vs. No Diet; Least Square Mean at follow up adjusted for the following covariates: baseline measure of the outcome measure, sex, and beta blocker usage
Statistical Analysis 2: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Test type: Superiority; p < 0.001, ANCOVA — Main effects analysis with Exercise vs. No Exercise; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Quality of Life
Description: Heart failure-specific quality of life was assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ) on a range 0-100; higher scores indicate better quality of life.
Time Frame: 20 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Exercise Training | Dietary Intervention | Attention Control | Diet and Exercise
Number analyzed (Participants) | 24 | 24 | 22 | 22
units on a scale | 71 [67 to 75] | 77 [73 to 81] | 69 [63 to 75] | 79 [75 to 84]
Statistical Analysis 1: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Test type: Superiority; p = 0.004, ANCOVA — Main effects analyses with Diet vs. No Diet; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Test type: Superiority; p = 0.43, ANCOVA — Main effects analysis for Exercise vs. No Exercise; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Body Composition
Description: Total Body Fat Mass and Total Non-bone Lean Mass via DEXA
Time Frame: 20 weeks
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Exercise Training | Dietary Intervention | Attention Control | Diet and Exercise
Number analyzed (Participants) | 24 | 24 | 22 | 22
kg
  Total Fat | 45 [43 to 47] | 42 [40 to 44] | 47 [45 to 49] | 40 [38 to 42]
  Total Non-Bone Lean | 52 [50 to 54] | 50 [50 to 50] | 53 [53 to 53] | 50 [48 to 52]
Statistical Analysis 1: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Total Body Fat Mass; Test type: Superiority; p < 0.001, ANCOVA — Main effects analyses with Diet vs. No Diet; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Total Body Fat Mass; Test type: Superiority; p = 0.001, ANCOVA — Main effects analysis of Exercise vs. No Exercise; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Total Non-Bone Lean Mass; Test type: Superiority; p < 0.001, ANCOVA — Main effects analyses with Diet vs. No Diet; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Total Non-Bone Lean Mass; Test type: Superiority; p = 0.25, ANCOVA — Main effects analysis for Exercise vs. No Exercise; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Thigh Muscle Composition
Description: Thigh Skeletal Muscle and Subcutaneous Fat via MRI
Time Frame: 20 weeks
Measure: Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Exercise Training | Dietary Intervention | Attention Control | Diet and Exercise
Number analyzed (Participants) | 24 | 24 | 22 | 22
cm^2
  Thigh Subcutaneous Fat | 155 [149 to 161] | 143 [137 to 149] | 164 [158 to 170] | 144 [138 to 150]
  Thigh Skeletal Muscle | 120 [118 to 122] | 115 [113 to 117] | 121 [117 to 125] | 114 [112 to 116]
Statistical Analysis 1: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Thigh Subcutaneous Fat; Test type: Superiority; p < 0.001, ANCOVA — Main effects analyses with Diet vs. No Diet; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Thigh Subcutaneous Fat; Test type: Superiority; p = 0.26, ANCOVA — Main effects analysis for Exercise vs. No Exercise; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Thigh Skeletal Muscle; Test type: Superiority; p < 0.001, ANCOVA — Main effects analyses with Diet vs. No Diet; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Exercise Training vs Dietary Intervention vs Attention Control vs Diet and Exercise; Thigh Skeletal Muscle; Test type: Superiority; p = 0.26, ANCOVA — Main effects analysis of Exercise vs. No Exercise; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Exercise Training | Dietary Intervention | Attention Control | Diet and Exercise
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/24 | 1/25 | 1/25
Other Adverse Events (participants affected / at risk) | 2/26 | 1/24 | 0/25 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise Training (N=26) | Dietary Intervention (N=24) | Attention Control (N=25) | Diet and Exercise (N=25)
Heart failure exacerbation (Cardiac disorders) | 0 | 0 | 0 | 1 (3)
Pancreatitis (Endocrine disorders) | 1 (1) | 0 | 0 | 0
Leg edema (Blood and lymphatic system disorders) | 0 | 0 | 1 (2) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise Training (N=26) | Dietary Intervention (N=24) | Attention Control (N=25) | Diet and Exercise (N=25)
Hypoglycemia (Endocrine disorders) | 0 | 1 (1) | 0 | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Stress fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0
Tendon tear (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No